CLINICAL TRIAL: NCT05368636
Title: Analyzing the Link Between Tongue Images and Gastric Cancer Cascade Response Using Artificial Intelligence Techniques
Brief Title: Combining Tongue and Gastric Cancer Cascade With Artificial Intelligence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, doctoral supervisor of Qilu Hospital gastroenterology department, Shandong University
Other Study IDs: 2022SDU-QILU-G001
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Artificial Intelligence; Tongue; Gastric Cancer
Keywords: Artificial Intelligence; tongue; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study combines artificial intelligence with tongue images, by collating and collecting tongue images and diagnostic and pathological results of gastroscopic diseases, mining and analysing the correlation between tongue images and OLGA, OLGIM stages, Correa sequences and constructing prediction models, to deeply investigate the relationship between tongue images and precancerous diseases, precancerous lesions and gastric cancer.

DETAILED DESCRIPTION:
Firstly, tongue pictures and patient information will be collected after the patient signed an informed consent form.

Secondly, after the patient undergoes gastroscopy, patient gastroscopy reports and pathology reports will be obtained.

Thirdly, the investigator will assess the patient's gastroscopy report for the Correa sequence of gastric cancer with OLGA and OLGIM staging.

Finally, the patient's tongue image, information and gastric cancer cascade response are matched to construct an artificial intelligence model and assess the quality of the model.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 40 and 80 years of age who are scheduled for gastroscopy.
* Patients all gave their informed consent and signed the informed consent form.

Exclusion Criteria:

* Persons with severe cardiac, cerebral, pulmonary or renal dysfunction or psychiatric disorders who are unable to participate in gastroscopy.
* Patients with previous surgical procedures on the gastrointestinal tract.
* Patients taking bismuth or other staining drugs.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 40-80 years who will undergo gastroscopy and fulfil the inclusion criteria who do not meet the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 3 years
  Sensitivity of artificial intelligence models Sensitivity = number of true positives / (number of true positives + number of false negatives) * 100%.
Specificity | 3 years
  Specificity of Artificial Intelligence Models Specificity = number of true negatives / (number of true negatives + number of false positives))*100%
Positive predictive values(PPV) | 3 years
  Positive predictive values from artificial intelligence models Positive predictive value = true positive / (true positive + false positive)*100%
Negative predictive values(NPV) | 3 years
  Negative predictive values for artificial intelligence models Negative predictive value = true negative / (true negative + false negative)*100%
AUC (95% CI) | 3 years
  area under the receiver operating characteristic curve (AUC)
Accuracy | 3 years
  Accuracy of artificial intelligence models Accuracy = (true positives + true negatives) / total number of subjects * 100%

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hosipital, Jinan, Shandong, China